CLINICAL TRIAL: NCT01217983
Title: Utility of Renal Biomarkers in Cirrhotic Patients
Brief Title: Utility of Renal Biomarkers in Cirrhosis
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Ponte Belen, Dr, University Hospital, Geneva
Other Study IDs: 10-056 Med 10-019; PRD 2010-I-15 (Other Grant/Funding Number: Projet de recherche et développement (PRD))
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Cirrhosis; Ascitis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum, urine and ascitis
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Evaluation of kidney function is critical in cirrhotic patients as there is a clear relationship between renal failure and prognosis. The investigators hypothesized that in this population new biomarkers of renal function could help in early detection of acute renal failure and in discrimination between renal and pre-renal causes. Finally the investigators hypothesized that such biomarkers could predict short-term outcome in this population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Known or suspected cirrhosis
* Suspected ascitis
* Informed consent signed

Exclusion Criteria:

* Proven multifocal hepatocellular carcinoma
* Acute gastric hemorrhage (active or < 2 weeks)
* Known end-stage renal disease or on dialysis before admission
* Recipients of kidney or liver transplants
* Transferred from another institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted for cirrhotic ascitis in the University Hospital of Geneva.
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Early detection of acute kidney injury in hospitalized cirrhotic patients with ascitis using new renal biomarkers | 30 days
  Acute kidney injury will be defined using RIFLE and AKIN criteria.

SECONDARY OUTCOMES:
Prediction of adverse clinical outcomes (Renal replacement therapy, transfer to ICU, all cause mortality). | 30 days
Discrimination between different type of AKI. | 30 days
Prediction of AKI developement using renal artery resistive indexes. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Belen Ponte, Md, Principal Investigator — Nephrology Division
Locations (1):
- University Hospital of Geneva, Geneva, Switzerland